CLINICAL TRIAL: NCT02499575
Title: Exparel Pericapsular Injection: A Prospective Evaluation of Postoperative Pain in Bunion Surgery, First Metatarsophalangeal Joint Fusion, and Cheilectomy
Brief Title: Pericapsular Exparel for Pain Relief in Bunionectomy and Related Procedures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical issues prevent efficient enrollment
Sponsor: OhioHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OH2-15-0005
Record Dates: First submitted 2015-07-02; First posted 2015-07-16 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2016-07

CONDITIONS: Bunion; Hallux Rigidus
Keywords: Exparel; bupivacaine; Hallux valgus deformity; bunionectomy
MeSH Terms: conditions — Bunion; Hallux Rigidus | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regional Block (Active Comparator): Group A patients will receive only a pre-operative adductor canal block with 10 mL 0.5% ropivacaine plus a popliteal block with 30 mL 0.5% ropivacaine (total block 40 mL/200 mg).
  Interventions: Drug: 0.5% ropivacaine
- Regional Block Plus Exparel (Experimental): Group B patients will receive the standard of care pre-operative adductor and popliteal block as described (40 mL/200 mg of 0.5% ropivacaine) in addition to a postoperative pericapsular injection of Exparel using 106 mg (8 mL, equivalent to 120 mg bupivacaine HCl), per the same total dose as provided in manufacturer recommendations.
  Interventions: Drug: 0.5% ropivacaine; Drug: Exparel

INTERVENTIONS:
Drug: 0.5% ropivacaine — Adductor block: 10 mL of 0.5% ropivacaine; popliteal block: 30 mL of 0.5% ropivacaine
  Other Names: ropivacaine
Drug: Exparel — 106 mg (8 mL, equivalent to 120 mg bupivacaine HCl)
  Other Names: Liposomal bupivacaine
  Arms: Regional Block Plus Exparel

SUMMARY:
Exparel is an FDA-approved local anesthetic (bupivacaine), in a long-release formulation. In this study the investigators plan to determine the ability of Exparel to control post-operative pain in common first metatarsophalangeal (MTP) joint procedures (bunion surgery, 1st MTP fusion, and cheilectomy).

DETAILED DESCRIPTION:
The investigators propose a prospective, randomized, single-blinded study of patients who are electing to undergo an outpatient first metatarsophalangeal (MTP) joint procedure (bunionectomy, 1st MTP fusion, or cheilectomy). As a standard, patients undergoing these procedures are given regional anesthesia (adductor canal block plus popliteal block). Patients are then given prescriptions for oral opioids to manage post-operative pain. The purpose of this study is to determine whether a single intrapopliteal administration of Exparel, in conjunction with the standard of care regional block, improves pain relief and therefore decreases use of post-operative opioids.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Undergoing distal or midshaft osteotomy for bunion correction, 1st MTP Fusion, or cheilectomy

Exclusion Criteria:

* Age less than 18
* Unable to read/write English
* Dementia, history of dementia, or other significant mental impairment that would, in the opinion of the investigator, impede patient self-reporting
* Weight <70 kg
* Allergy to local anesthetics
* History of long-acting opioid use or opioid tolerance (any patient receiving at least 30 mg of oxycodone or equivalent per day (e.g., 6 tabs of Percocet 5/325 mg) regularly for approximately 7 days or more OR who require increased analgesic doses for a period long enough to develop tolerance to the effects of the opioid including analgesia and sedation)
* Any history of opioid misuse, illicit or prescription
* Prior MTP joint correction on the surgical limb
* Midfoot and hindfoot procedures performed concurrently, on the same day
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hyer, DPM, Principal Investigator — OhioHealth
Locations (2):
- United States (2):
  - Grant Medical Center, Columbus, Ohio
  - Orthopedic Foot and Ankle Center, Westerville, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regional Block | Regional Block Plus Exparel
Started | 1 | 1
Completed | 1 | 0
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regional Block | Regional Block Plus Exparel | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Customized [Number; unit: years]
  Age | 62 |  | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use as Measured by Questionnaire
Description: Compare time to first opioid use over 72 hours between groups
Time Frame: Daily through the third day (72 hours) post-surgery
Measure: Number; unit: hours
Arm/Group | Regional Block | Regional Block Plus Exparel
Number analyzed (Participants) | 1 | 0
hours | 6 |

2. Primary Outcome: Total Opioid Use as Measured by Questionnaire
Description: Compare total opioid use (reported as total morphine equivalents) over 72 hours between groups.
Time Frame: Daily through the third day (72 hours) post-surgery
Measure: Number; unit: morphine equivalents
Arm/Group | Regional Block | Regional Block Plus Exparel
Number analyzed (Participants) | 1 | 0
morphine equivalents | 18 |

3. Secondary Outcome: Pain Relief Measured by Defense and Veterans Pain Scale
Description: Evaluate patient-reported pain scores (scale of 0 (no pain) - 10 (worst pain)) at 0, 6, 12, 24, 36, 48, 60, and 72 hours following surgery
Time Frame: Through 72 hours post-surgery (0, 6, 12, 24, 36, 48, 60, and 72 hours post-surgery)
Measure: Number; unit: units on scale of 0 -10
Arm/Group | Regional Block | Regional Block Plus Exparel
Number analyzed (Participants) | 1 | 0
units on scale of 0 -10
  Pain score time 0 | 0 |
  Pain score time 6hrs | 3 |
  Pain score time 12hrs | 3 |
  Pain score time 24hrs | 2 |
  Pain score time 36hrs | 3 |
  Pain score time 48hrs | 3 |
  Pain score time 60hrs | 2 |
  Pain score time 72hrs | 2 |

ADVERSE EVENTS:
Time Frame: up to 30 days
Arm/Group | Regional Block | Regional Block Plus Exparel
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No